CLINICAL TRIAL: NCT01409954
Title: Defining the Osteogenic Potential of Mesenchymal Stem Cells and Their Progenitors During Spinal Decompression and Posterolateral Lumbar Fusion
Brief Title: Collecting Bone Graft During Spinal Decompression and Posterolateral Lumbar Fusion to Better Define Bone Making Cells
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brandon Lawrence, M.D., University of Utah
Other Study IDs: 46970
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pseudarthrosis After Fusion or Arthrodesis
Keywords: Fusion; Spine; Decompression; Pseudarthrosis; bone harvest; Instrumented posterolateral fusion
MeSH Terms: conditions — Ankylosis; Pseudarthrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aliquots of bone marrow aspirates and bone fragments
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal decompression: Spinal decompression with an instrumented posterolateral fusion

SUMMARY:
The purpose of this study is to improve fusion (bony healing) techniques and improve patient recovery by identifying cells in your body that make bone. Patients with spine problems often need surgeries that include fusion (bony healing) of vertebrae (bones in your back) together in order to hold the bones steady allowing them to heal together (fusion). If the vertebrae (back bones) fail to heal together, which occurs about 10-15% of the time, it can result in a slower recovery and may require revision (another) surgery. By using a small portion of the graft taken during surgery the investigators hope to define the cells that make bone most efficiently. This will help reduce the need for revision surgeries and improve patient recovery.

DETAILED DESCRIPTION:
This study requests using your additional bone tissue (the extra tissue not needed after your back surgery is complete).

This tissue will be measured for total volume (amount), labeled with your age, gender, date and time the tissue was removed (date and time of surgery), and taken to a lab for analysis. You will not be billed for the collection of your additional tissue or the lab analysis. All routine procedures (surgery and all follow-up care relating to your back surgery) will still be paid for by you or your insurance.

Once your extra tissue sample has been collected, measured, labeled, and sent to the lab for testing, no further participation is required from you in this research study. The investigators will use your sample in our research to enhance bone healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo spinal decompression with an instrumented posterolateral fusion

Exclusion Criteria:

* Patients not undergoing spinal decompression with an instrumented posterolateral fusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialty clinic, University of Utah Orthopaedic Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Osteogenic Potential of Mesenchymal Stem Cells | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Lawrence, MD, Principal Investigator — University of Utah Department of Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States